CLINICAL TRIAL: NCT05327036
Title: The Effect of Single Umbilical Artery Caused by Umbilical Artery Embolism on Pregnancy Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2022-07-202
Record Dates: First submitted 2022-03-30; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Umbilical Artery Embolism,Single Umbilical Artery,Pregnancy Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- pregnant women with Single Umbilical Artery: pregnant women with Single Umbilical Artery
  Interventions: Other: collect information about all participants
- pregnant women with Umbilical Artery Embolism: pregnant women with Umbilical Artery Embolism
  Interventions: Other: collect information about all participants
- Normal pregnant women: Normal pregnant women without pregnancy complications
  Interventions: Other: collect information about all participants

INTERVENTIONS:
Other: collect information about all participants — collect information On age,pregnancy history,Height, weight,Gestational weeks of umbilical artery embolism,Gestational week of delivery, mode of delivery, newborn birth weight, birth height, Apgar score, umbilical cord length, umbilical cord placental insertion point, placental weight, pregnancy complications, coagulation function,after obtaining the consent of all participants.

SUMMARY:
To investigate the relationship between single umbilical artery caused by umbilical artery embolism and pregnancy outcome , and to provide evidence-based evidence for peripartum health care of pregnant women with umbilical artery embolism.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 ~ 34years old
* B-ultrasound first showed double umbilical artery, then single umbilical artery or pregnant women with umbilical artery embolism supported by intrapartum and postpartum pathology.
* B-ultrasound of prenatal examination showed a single umbilical artery, and prenatal and postpartum pathology showed pregnant women with a single umbilical artery.

Exclusion Criteria:

* The fetus has extracardiac malformation and aneuploid deformity

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligible participants is female.
Study Population: The participants include women with pregnancy meeting the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Gestational week of delivery | 32 weeks to 40 weeks gestation
  The gestational age of delivery is determined according to the last menstruation and ultrasonic diagnosis.
mode of delivery | 32 weeks to 40 weeks gestation
  The mode of delivery including vaginal delivery and cesarean section, is determined by the exact condition of pregnancy.
newborn birth weight | 32 weeks to 40 weeks gestation
  Newborn weight is measured immediately after birth.
birth height | 32 weeks to 40 weeks gestation
  Birth height is measured immediately after birth.
Apgar score | 32 weeks to 40 weeks gestation
  Apgar score is assessed at 1 min and 5 minute after birth.

SECONDARY OUTCOMES:
coagulation function | 32 weeks to 40 weeks gestation
  Coagulation function including prothrombin time and activated partial thromboplastin time is measured just before delivery.
placental weight | 32 weeks to 40 weeks gestation
  Placental weight is measured after delivery of the placenta.
umbilical cord placental insertion point | 32 weeks to 40 weeks gestation
  The placenta is observed after delivery to determine the insertion point of the umbilical cord in placenta.
umbilical cord length | 32 weeks to 40 weeks gestation
  Umbilical cord length is measured after delivery of the neonate.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Hua, Study Director — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- department of obstetrics of Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China